CLINICAL TRIAL: NCT03694106
Title: Feasility Pilot of T.E.A.M. Psychotherapy Using Electronic Capture of Before and After Therapy Measures.
Brief Title: T.E.A.M. Feasibility and Efficacy Study 2.0
Acronym: TEAM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Feeling Good Institute (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Alex Clarke, Director of Research and Development, Feeling Good Institute
Other Study IDs: 41809
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: TEAM PSYCHOTHERAPY — Patients data will be collected from the first to the final psychotherapy session as performed normally by TEAM trained clinicians. The treatment-as-usual includes therapy sessions of 50 to 110minutes long, typically once or twice per week for an average of 8-12 sessions. Treatment as usual by these clinicians includes the use of psychological symptoms survey immediately before and after each psychotherapy session. Typically patients will fill out these surveys in the clinic's waiting area before and after each session.

SUMMARY:
T.E.A.M. psychotherapy was developed by one of the founders of cognitive therapy, David Burns and builds on traditional CBT with an emphasis on T = Testing, E = Empathy, A = Agenda Setting (assessing and building motivation) and M = Methods (including cognitive and behavioral methods). Because TEAM therapy is a data-driven therapy, its delivery hinges on the use of symptom measures and measures of the therapeutic alliance at every session with every patient. These measures are now available for collection thru computerized forms, making their collection and review considerably more accessible and efficient for the patient and therapist.

The following hypotheses will be tested:

1. TEAM psychotherapy using computerized measurement collection is safe and feasible.
2. TEAM psychotherapy using computerized measurement collection shows evidence of efficacy by exploratory non inferiority testing compared to benchmark studies with similar psychotherapeutic modalities
3. Evidence for efficacy is strong enough to justify pursuit of an experimental randomized controlled clinical trial of TEAM therapy for major depressive disorder versus treatment as usual.

DETAILED DESCRIPTION:
A gap currently exists between the technology available for collecting psychotherapy data and the application of this technology to psychotherapeutic settings to enhance treatment outcomes. A novel integration of Cognitive Behavior Therapy (CBT) informed psychotherapy and digitized data collection systems called T.E.A.M. therapy exists that bridges this gap and has yet to be tested. The purpose of this study is to explore whether TEAM CBT appears safe and feasible and has results similar to comparable and similar benchmark studies. This outcome will provide pilot data and a rationale for whether to pursue a separate randomized controlled trial in the future. We will compare the results of TEAM therapy using electronic data collection to similar psychotherapeutic treatments for common psychiatric problems such as depression, anxiety, relationship conflicts and maladaptive behaviors. We will also explore the data for its use in predictive modeling. This study is part of a wider goal of developing best practices in dissemination of standardized measurement based psychotherapies that are effective and use technology via computerized delivery systems guided by therapists. It is hoped that with computer based measurement systems for psychotherapy, more accurate and frequent information for therapists is available to modify earlier and more effectively their approaches. The measurement based systems will also allow performance by psychotherapists to be measured accurately and enable a type of machine based learning environment with feedback systems in place to improve providers' patient care in a more precise and personalized way.

ELIGIBILITY:
Inclusion Criteria:

* 1. Cognitive functioning at a level and ability to use an electronic tool. 2. Demonstration of decisional capacity in order to participate in psychotherapy.

Exclusion Criteria:

1. Under age 18 3. Providers: not TEAM certified at a level 3 or above 2. Patients: Non-fluent English speakers. The tool for now is only available in English

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Receiving TEAM therapy from Level 4 or above therapist.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
NIH PROMIS 4 item depression questionnaire | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Maor Katz, MD, Principal Investigator — Feeling Good Institute; Alex Clarke, MD, Principal Investigator — Feeling Good Institute
Locations (1):
- Feeling Good Institute, Mountain View, California, United States

IPD SHARING:
Plan to Share IPD: Undecided